CLINICAL TRIAL: NCT05747768
Title: A Clinical Study to Evaluate the Pharmacokinetics of Microdose Midazolam, Dabigatran, Pitavastatin, Atorvastatin and Rosuvastatin in Healthy Volunteers and Renal Impairment Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dongyang Liu, Researcher, Peking University Third Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DCTC-IIR202229
Record Dates: First submitted 2023-02-06; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Midazolam; Dabigatran; pitavastatin; Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy Volunteers (Experimental): Healthy volunteer received drug combinations（10 µg midazolam, 375 µg dabigatran etexilate, 10 µg pitavastatin, 50 µg rosuvastatin, and 100 µg atorvastatin） on an empty stomach
  Interventions: Drug: Midazolam, dabigatran etexilate, pitavastatin, rosuvastatin and atorvastatin
- Patients with mild-to-moderate renal impairment (Experimental): Patients with mild-to-moderate renal impairment received drug combinations（10 µg midazolam, 375 µg dabigatran etexilate, 10 µg pitavastatin, 50 µg rosuvastatin, and 100 µg atorvastatin） on an empty stomach
  Interventions: Drug: Midazolam, dabigatran etexilate, pitavastatin, rosuvastatin and atorvastatin
- Patients with moderate to severe renal impairment (Experimental): Patients with moderate to severe renal impairment received drug combinations（10 µg midazolam, 375 µg dabigatran etexilate, 10 µg pitavastatin, 50 µg rosuvastatin, and 100 µg atorvastatin） on an empty stomach
  Interventions: Drug: Midazolam, dabigatran etexilate, pitavastatin, rosuvastatin and atorvastatin
- Patients with severe renal impairment (Experimental): Patients with severe renal impairment received drug combinations（10 µg midazolam, 375 µg dabigatran etexilate, 10 µg pitavastatin, 50 µg rosuvastatin, and 100 µg atorvastatin） on an empty stomach
  Interventions: Drug: Midazolam, dabigatran etexilate, pitavastatin, rosuvastatin and atorvastatin
- Patients with end-stage renal disease (Experimental): Patients with end-stage renal disease received drug combinations（10 µg midazolam, 375 µg dabigatran etexilate, 10 µg pitavastatin, 50 µg rosuvastatin, and 100 µg atorvastatin） on an empty stomach
  Interventions: Drug: Midazolam, dabigatran etexilate, pitavastatin, rosuvastatin and atorvastatin

INTERVENTIONS:
Drug: Midazolam, dabigatran etexilate, pitavastatin, rosuvastatin and atorvastatin — Midazolam, dabigatran etexilate, pitavastatin, rosuvastatin and atorvastatin were provided by the Department of Pharmacy, Peking University Third Hospital, and were dissolved and mixed with normal saline respectively, and the mixing process needed to be fully stirred. Then, according to the concentration of the drug mixed solution, the corresponding volume of mixed solution was given to achieve the dosage of 10 μg midazolam, 375 μg dabigatran etexilate, 10 μg pitavastatin, 50 μg rosuvastatin and 100 μg atorvastatin. In order to avoid the food effect, the test drugs were administered on an empty stomach on the administration day in this experiment.

SUMMARY:
1. To explore the functional changes of P-gp, CYP3A4, OATP1B and BCRP in Chinese people with renal impairment;
2. To explore the effect of dialysis on the functional changes of P-gp, CYP3A4, OATP1B and BCRP in patients with end-stage renal disease;
3. Validation of urotoxic molecules as possible biomarkers that can assess intestinal P-gp function.

ELIGIBILITY:
Inclusion Criteria:

All participants:

1. male or female , Chinese (individuals have Chinese descent) subjects, Age between 18-65 (include) with the ability of cognizance;
2. body mass index (BMI) of 18.5 to 24 kg/m2 for all participants ; body weight for male >50 kg; a total body weight for female >45 kg;
3. female must be non-pregnant, non-breast feeding and if she is reproductive potential: must agree to use (and/have their partner use) effective methods of birth control beginning at screening ,throughout the study and until 6 months after last dosing of study drug;
4. is a non-smoker or moderate smoker (≤20 cigarettes/day or the equivalent);
5. signed the Inform Consent Form , fully understood the trial conduction and comply with the requirement of the research;

Participants with mild to moderate , moderate to severe , severe renal impairment or end stage renal disease:

1. has a clinical diagnosis of renal impairment and meets the protocol-specified renal impairment function qualifications at screening;
2. with the classification of KDIGO (Kidney Disease Improving Global Outcomes ), the mild to moderate renal impairment patients have eGFR between 45 to 90(include) mL/min/1.73m2 based on MDRD (Modification of Diet in Renal Disease Study) equation, without dialysis before;
3. with the classification of KDIGO (Kidney Disease Improving Global Outcomes ), the moderate to severe renal impairment patients have eGFR between 30 to 44(include) mL/min/1.73m2 based on MDRD(Modification of Diet in Renal Disease Study) equation, without dialysis before;
4. with the classification of KDIGO (Kidney Disease Improving Global Outcomes ), The moderate to severe renal impairment patients have eGFR between 15 to 29(include) mL/min/1.73m2 based on MDRD(Modification of Diet in Renal Disease Study) equation, without dialysis before;
5. with the classification of KDIGO (Kidney Disease Improving Global Outcomes ), The end stage renal disease patients have eGFR below 15 (include) mL/min/1.73m2 based on MDRD(Modification of Diet in Renal Disease Study) equation, with dialysis therapy;
6. participants with mild to moderate , moderate to severe , severe renal impairment or end stage renal disease: With stable renal function lasted for three months before first oral dose ; the shrinkage of eGFR be within 30%;

Healthy participants ,besides:

1. has baseline eGFR ≥ 90 mL/min based on MDRD (Modification of Diet in Renal Disease Study) equation;
2. is judged to be in good health based on medical history, physical examination, vital signs and laboratory safety tests, without clinically significant laboratory abnormalities.

Exclusion Criteria:

1. is mentally or legally incapacitated at the time of the screening visit or expected during the conduct of the study;
2. history of stroke, chronic seizures, or major neurological disorders;
3. history of malignant neoplastic disease;
4. history or presence of alcoholism or drug abuse within the past 6 months;
5. history of hypersensitive reaction or allergic to study drug (including midazolam, dabigatran Etexilate, pitavastatin, atorvastatin, rosuvastatin), only if with researchers permission;
6. blood donation within the past 4 weeks or lost more than 500 mL blood before screening;
7. apheresis within the past 8 weeks before screening;
8. take weak/moderate inhibiters or inducers of CYP3A/BCRP/OATP1B/P-gp within 14 days before screening, including but not limited to: clarithromycin, boceprevir, cobicistatdanoprevir, grapefruit juice, indinavir, ketoconazole, telaprevir, paritaprevir, Telithromycin, troleandomycin, voriconazole, nafazodone, Idelalisib, nelfinavir, fluconazole, aprepitant, ciprofloxacin, conivaptan , crizotinib, cyclosporin A, diltiazem, fluvoxamine, imatinib, tofisopam, atazanavir, erythromycingemfibrozilsimepreviramiodarone, carvedilol, itraconazole, lapatinib, lopinavir, ritonavir, propafenone, quinidine, ranolazine, saquinavir, telaprevir, verapamil, tipranavir, curcumin, Eltrombopag, phenytoin, rifampicin, apalutamide, carbamazepine, St. John's Wort, mitotan, enzalutamide, bosentan, efavirenz, primidone, phenobarbital;
9. intolerance of venous blood collection;
10. history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, immunological, respiratory, or genitourinary abnormalities or diseases, include cancer, traumatic brain injury, persistent viral infection, rheumatoid arthritis, inflammatory bowel disease, NAFLD, Liver cirrhosis, HIV, Hyperthyreosis, Cushing syndrome, Parkinson or has a history of Parkinson in his family;
11. history of myocardial infarction, cerebral stroke, cerebral infarction within 3 months;
12. history of gastrointestinal diseases: irritable bowel syndrome, enteric bacterial overgrowth syndrome, gastroesophageal reflux disease, Gallstones, coeliac disease, Crohn disease, Ulcerative Colitis, active peptic ulcers;
13. subjects who test positive at screening for human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B surface antigen (HbsAg), and syphilis;

Participants with mild to moderate, moderate to severe, severe renal impairment or end stage renal disease,exclusion criteria are appended below:

1. history of renal transplant or nephrectomy;
2. presence of uncontrolled type 2 diabetes mellitus (T2DM), a history of type 1 diabetes or ketoacidosis;
3. participants with rapid fluctuation of renal function according to previous laboratory examination; or have been diagnosed of renal stenosis. The definition of rapid fluctuation of renal function refers to the fluctuation of eGFR greater than 30% within 3 months after the examination. If no historical measurements are available, two examinations will be used to demonstrate stability: fluctuation of eGFR less than 30% between two consecutive examinations within 3 months before screening;

Healthy participants ,exclusion criteria are appended below:

1.presence of hypoglycemia, glucose intolerance,uncontrolled type 2 diabetes mellitus (T2DM) or ketoacidosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
plasma concentration | Baseline and within 24 hours after administration
dialysate concentration | 1 day

SECONDARY OUTCOMES:
biomarker concentration | Baseline and within 24 hours after administration
urine concentration | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China